CLINICAL TRIAL: NCT01400815
Title: A Prospective, Double-blind, Randomized, Active Controlled, Parallel Group, Multicenter Phase II Clinical Trial to Evaluate the Effectiveness of X-22 as a Smoking Cessation Aid
Brief Title: Randomized Trial to Evaluate the Effectiveness of X-22 as a Smoking Cessation Aid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: 22nd Century Limited, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: X-22-201
Record Dates: First submitted 2011-07-19; First posted 2011-07-22 (Estimated); Results first posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-10

CONDITIONS: Smoking Cessation
Keywords: smoking; smoking cessation; quitting smoking
MeSH Terms: conditions — Smoking Cessation; Smoking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- X-22 Smoking Cessation Product (Experimental): The X-22 Smoking Cessation Product is a tobacco-based (botanical) medical product consisting of very low nicotine (VLN) cigarettes.
  Interventions: Drug: X-22 Smoking Cessation Product
- Active Control Cigarette (Active Comparator): The Active Control cigarette is identical to the X-22 cigarette except for the tobacco, which has a nicotine content similar to that of a conventional "light" cigarette.
  Interventions: Drug: Active Control Cigarettes

INTERVENTIONS:
Drug: X-22 Smoking Cessation Product — The X-22 Smoking Cessation Product is a tobacco-based (botanical) medical product consisting of very low nicotine (VLN) cigarettes.
  Subjects will be allowed to smoke as much as desired throughout the 6-week treatment period.
  Arms: X-22 Smoking Cessation Product
Drug: Active Control Cigarettes — The Active Control cigarette is identical to the X-22 cigarette except for the tobacco, which has a nicotine content similar to that of a conventional "light" cigarette.
  Subjects will be allowed to smoke as much as desired throughout the 6-week treatment period.
  Arms: Active Control Cigarette

SUMMARY:
A randomized, active controlled clinical trial in which a total of 216 healthy smokers will be enrolled and followed over approximately 19 weeks.

The trial will evaluate the efficacy and safety of using X-22 as a smoking cessation aid.

Healthy smokers who plan to quit smoking will be screened for eligibility. Subjects will be randomized in a 1:1 ratio to 1 of the 2 treatment arms:

* Group 1: X-22 Cigarettes (very low nicotine)
* Group 2: Active Control Cigarettes The randomization will be stratified by gender. Efficacy will be assessed by analysis of cigarette consumption using self-report diaries and measurement of exhaled carbon monoxide (CO) and cotinine concentrations.

Safety will be assessed by evaluation of adverse events, physical examinations, clinical laboratory tests, and measurement of heart rate, blood pressure, and body weight at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible for participation in this study.

  1. Subjects must be considered by the investigator to be in general good health and between 18 and 65 years of age, inclusive.
  2. Subjects must have a history of smoking at least 10 cigarettes per day for at least 1 year, with less than 3 months of abstinence during the past year, and a continuous smoking history for at least 3 months prior to study entry.
  3. Subjects must indicate that they plan to quit smoking within the next 3 months.
  4. Subjects must have a CO measurement of ≥ 10 ppm at screening and baseline (Visit 1 and Visit 2).
  5. Subjects must be willing and able to return for scheduled follow-up examinations for a total of 5 months.
  6. Female subjects must have been postmenopausal for the previous 6 months or be surgically sterile, or must have a negative pregnancy test and use one of the following acceptable methods of birth control for the duration of the study and for at least 3 months prior to screening:
* abstinence, meaning a total lack of sexual activity,
* oral contraceptives ("the pill"),
* contraceptive injections,
* intrauterine device,
* double-barrier method (diaphragm or condom plus spermicidal cream),
* contraceptive patch, hormonal implant, hormonal vaginal ring, or
* male partner sterilization at least 3 months prior to screening. 7. Subjects must sign and be given a copy of the written Informed Consent form. 8. Subjects must be able to read, understand and complete the questionnaires independently.

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria are not to be enrolled in this study.

  1. Subjects who have a household member who is already enrolled in this trial.
  2. Subjects who have attempted to quit smoking using one or more FDA-approved smoking cessation products (eg, nicotine replacement therapy [NRT] including nicotine gum, nicotine lozenges, nicotine patches, nicotine nasal spray, or nicotine inhaler; Zyban [bupropion]; or Chantix [varenicline]) for longer than 1 week in the past 3 months.
  3. Subjects who have been enrolled in another structured smoking cessation program (e.g., behavioral modification, hypnosis, acupuncture, or other alternative therapies) in the last 30 days.
  4. Subjects who have been in another smoking cessation trial in the past 6 months.
  5. Subjects who regularly use (greater than once per month) tobacco-based products other than cigarettes (eg, chew, snuff, snus, shisha, etc.).
  6. Subjects with a history of coronary artery disease, myocardial infarction, stroke, chronic obstructive pulmonary disease, or other significant pulmonary diseases. Controlled hypertensive subjects and mild asthmatics whose disease is controlled only with an as-needed inhaled beta agonist are acceptable.
  7. Subjects with a history of cancer within the past 60 months other than basal cell carcinoma.
  8. Subjects with a history of thromboembolic disease or taking warfin or any other anticoagulant, or anti-platelet drug such as clopidogrel (Plavix®) or pentoxifylline (Trental®). Low dose aspirin therapy is acceptable.
  9. Subjects with screening laboratory abnormalities that are considered by the investigator to be clinically significant.
  10. Subjects with a body mass index (BMI) >35.
  11. Subjects with poorly controlled diabetes or insulin-dependent diabetes.
  12. Subjects with other known serious pathophysiology or topical or systemic disorders of any kind that would confound the results of the study.
  13. Subjects with screening ECG abnormalities that are considered by the investigator to be clinically significant.
  14. Subjects who have used any illegal drug in the past 3 months.
  15. Subjects who have a positive urine drug screening result.
  16. Subjects who are pregnant or lactating, or who plan to become pregnant during the course of the study.
  17. Subjects participating in any other clinical trial of an investigational drug or device during the time of this clinical investigation or within 30 days prior to Screening visit.
  18. Subjects taking anti-depressants, anti-psychotics, clonidine, or any of the classes of drugs listed in the RapidCHECK® 12 Panel in the last 60 days (see Section 12.1.1).
  19. Subjects with systolic blood pressure over 140 mmHg and/or diastolic blood pressure over 90 mmHg.
  20. Subjects consuming an average of 3 or more drinks of alcohol per day.
  21. Subjects consuming greater than an average of 2 packs of cigarettes per day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Benchmark Research Sacramento, Sacramento, California
  - Benchmark Research New Orleans, Metairie, Louisiana
  - Benchmark Research Austin, Austin, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- X-22 Smoking Cessation Product: The X-22 Smoking Cessation Product is a tobacco-based (botanical) medical product consisting of very low nicotine (VLN) cigarettes.
  X-22 Smoking Cessation Product: The X-22 Smoking Cessation Product is a tobacco-based (botanical) medical product consisting of very low nicotine (VLN) cigarettes.
  Subjects will be allowed to smoke as much as desired throughout the 6-week treatment period.
- Active Control Cigarette: The Active Control cigarette is identical to the X-22 cigarette except for the tobacco, which has a nicotine content similar to that of a conventional "light" cigarette.
  Active Control Cigarettes: The Active Control cigarette is identical to the X-22 cigarette except for the tobacco, which has a nicotine content similar to that of a conventional "light" cigarette.
  Subjects will be allowed to smoke as much as desired throughout the 6-week treatment period.
Period: Overall Study
Arm/Group | X-22 Smoking Cessation Product | Active Control Cigarette
Started | 118 | 116
Completed | 80 | 95
Not Completed | 38 | 21
Not completed — Adverse Event | 3 | 0
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 18 | 11
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 15 | 8
Not completed — Subject in jail | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | X-22 Smoking Cessation Product | Active Control Cigarette | Total
Number analyzed (Participants) | 118 | 116 | 234
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.1 (11.0) | 41.8 (11.2) | 41.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 52 | 106
  Male | 64 | 64 | 128
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 26 | 33 | 59
  White | 88 | 81 | 169
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Efficacy - 4 Weeks of Continuous Abstinence From Smoking Cigarettes
Description: The primary efficacy measurement is the number of subjects with 4 weeks of continuous abstinence from smoking cigarettes (Weeks 7-10), as assessed by subject diary and confirmed by exhaled carbon monoxide (CO), after treatment termination, at Visits 6 and 7.
  A responder: did not smoke and had less than 10 ppm exhaled CO.
Time Frame: Weeks 7 and 9 = telephone call, Week 8 = visit 6 and Week 10 = visit 7
Population: intent to treat (ITT) population
Measure: Count of Participants; unit: Participants
Arm/Group | X-22 Smoking Cessation Product | Active Control Cigarette
Number analyzed (Participants) | 118 | 116
Participants
  Week 8 - No Cigarettes Smoked per Diary (Weeks 7 and 8) | 14 | 14
  Week 8 - Exhaled CO <= 10ppm | 32 | 36
  Week 8 responder | 14 | 11
  Week 10 - No Cigarettes Smoked per Diary (Weeks 9 and 10) | 16 | 18
  Week 10 - Exhaled CO <= 10ppm | 38 | 30
  Week 10 responder | 16 | 13
  Overall Responder | 13 | 10

ADVERSE EVENTS:
Arm/Group | X-22 Smoking Cessation Product | Active Control Cigarette
All-Cause Mortality (participants affected / at risk) | 0/118 | 1/116
Serious Adverse Events (participants affected / at risk) | 5/118 | 1/116
Other Adverse Events (participants affected / at risk) | 60/118 | 58/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | X-22 Smoking Cessation Product (N=118) | Active Control Cigarette (N=116)
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic coma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | X-22 Smoking Cessation Product (N=118) | Active Control Cigarette (N=116)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Astigmatism (Eye disorders) | 1 (1) | 0 (0)
Dark circles under eyes (Eye disorders) | 1 (1) | 0 (0)
Myopia (Eye disorders) | 1 (1) | 0 (0)
Retinal disorder (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oral Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 1 (1)
Irritability (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 2 (2) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 20 (20) | 17 (17)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 3 (3)
Tooth infection (Infections and infestations) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Varicella (Infections and infestations) | 1 (1) | 0 (0)
Ear Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Laceration (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic coma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood carbon monoxide increased (Investigations) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 1 (1) | 1 (1)
Blood pressure increased (Investigations) | 1 (1) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 1 (1)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Red blood cell count decreased (Investigations) | 0 (0) | 1 (1)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 8 (8)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1) | 1 (1)
VIIth nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0)
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 7 (7)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI's have a general obligation of confidentiality, which extends to the study results and data procured under the study. There are exceptions to this obligation of confidentiality, which include the disclosure of study information and results in connection with publication and is necessary for the medical care of a study subject.